CLINICAL TRIAL: NCT01712659
Title: Phase I/II Trial Evaluating the Safety and Efficacy of Ruxolitinib in Subjects With Smoldering and Chronic Adult T-cell Leukemia (ATL)
Brief Title: Ruxolitinib for Adult T-Cell Leukemia
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The adult T-cell leukemia (ATL) research program was terminated after the death of the T-cell malignancy group Lead investigator.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Kevin Conlon, MD, Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 130006; 13-C-0006
Record Dates: First submitted 2012-10-20; First posted 2012-10-23 (Estimated); Results first posted 2023-01-10 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2022-12

CONDITIONS: T Cell Leukemia, Adult; Leukemia, Adult T-Cell; T Cell Leukemia, HTLV I Associated
Keywords: JAK 1/2; Human T-Cell Lymphotropic Virus 1; HTLV-1; Janus Kinase Inhibitor
MeSH Terms: conditions — Leukemia-Lymphoma, Adult T-Cell; Leukemia, T-Cell | interventions — ruxolitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Original Phase II Standard Ruxolitinib dose cohort (Experimental): Ruxolitinib 20 mg orally twice daily for 28 days. Subjects may continue to receive treatment until progressive disease (PD) or unacceptable toxicity.
  Interventions: Drug: Ruxolitinib
- 2- Phase 1 Dose Escalation cohorts (Experimental): Dose level 1: Ruxolitinib 30 mg orally twice daily for 28 days to determine the maximum tolerated dose (MTD). Subjects may continue to receive treatment until progressive disease (PD) or dose limiting toxicity (DLT) or unacceptable toxicity.
  Dose level 2: Ruxolitinib: Ruxolitinib 40 mg orally twice daily for 28 days to determine the maximum tolerated dose (MTD). Subjects may continue to receive treatment until progressive disease (PD) or dose limiting toxicity (DLT) or unacceptable toxicity.
  Dose level 3: Ruxolitinib: Ruxolitinib 50 mg orally twice daily for 28 days to determine the maximum tolerated dose (MTD). Subjects may continue to receive treatment until progressive disease (PD) or dose limiting toxicity (DLT) or unacceptable toxicity.
  Interventions: Drug: Ruxolitinib
- 3- Phase 1 Dose Expansion Cohort (Experimental): Ruxolitinib at the maximum tolerated dose (MTD) or the maximum administered dose (MAD) defined in the phase 1 dose escalation cohorts. Subjects may continue to receive treatment until progressive disease (PD) or unacceptable toxicity.
  Interventions: Drug: Ruxolitinib

INTERVENTIONS:
Drug: Ruxolitinib — Ruxolitinib 20 mg orally twice daily for 28 days. Subjects may continue to receive treatment until progressive disease (PD) or unacceptable toxicity.
  Other Names: Jakafi
  Arms: 3- Phase 1 Dose Expansion Cohort; Original Phase II Standard Ruxolitinib dose cohort
Drug: Ruxolitinib — Ruxolitinib 30 mg orally twice daily for 28 days to determine the maximum tolerated dose (MTD). Subjects may continue to receive treatment until progressive disease (PD) or dose limiting toxicity (DLT) or unacceptable toxicity.
  Other Names: Jakafi
  Arms: 2- Phase 1 Dose Escalation cohorts
Drug: Ruxolitinib — Ruxolitinib: Ruxolitinib 40 mg orally twice daily for 28 days to determine the maximum tolerated dose (MTD). Subjects may continue to receive treatment until progressive disease (PD) or dose limiting toxicity (DLT) or unacceptable toxicity.
  Other Names: Jakafi
  Arms: 2- Phase 1 Dose Escalation cohorts
Drug: Ruxolitinib — Ruxolitinib 50 mg orally twice daily for 28 days to determine the maximum tolerated dose (MTD). Subjects may continue to receive treatment until progressive disease (PD) or dose limiting toxicity (DLT) or unacceptable toxicity.
  Other Names: Jakafi
  Arms: 2- Phase 1 Dose Escalation cohorts

SUMMARY:
Background:

* The human T-cell leukemia virus 1 (HTLV-1) causes adult T-cell leukemia (ATL). Infection does not immediately cause ATL, but it can develop over time. ATL is a rare and aggressive type of cancer that disrupts the body's ability to control the HTLV-1 virus. Infected T lymphocytes that are transformed by HTLV-1 into malignant ATL cell have constitutively activated Interleukin-2 (IL-2), IL-9 and IL-15 production pathways that function as autocrine and paracrine stimulators of these cells by stimulating these cells through the Janus Kinase (JAK) 1 and 3/Signal transducer and activator of transcription 5 (STAT5) pathways.
* Ruxolitinib is a drug that has been approved to treat bone marrow disorders. Ruxolitinib is a tyrosine kinase inhibitor that disrupts signaling through the JAK 1 and 2/STAT3 and 5 pathways and have potential as a treatment for ATL. Researchers want to see if ruxolitinib can be a safe and effective treatment for ATL.
* Initially this trial was designed as a single dose level phase II trial with ruxolitinib given at the dose approved for the treatment of primary myelofibrosis, post-polycythemia vera myelofibrosis and post-essential thrombocythemia myelofibrosis.
* Clinical and correlative laboratory data demonstrated limited inhibition and impact on the subject's disease with the standard 20 mg twice daily dose. Given that the manufacturers of ruxolitinib had safety data for administering ruxolitinib to normal healthy volunteers at doses up to 50 mg twice or 100 mg once daily, the trial was reconfigured as a phase I dose escalation trial giving these higher doses on the twice daily schedule

Objectives:

Initial Phase II design:

* Define clinical or objective response rate for the 20 mg twice daily dose of Ruxolitinib.
* Define safety profile, Time to progression and survival time.

Subsequent Phase I dose escalation with expansion cohort treated at the MTD or MAD:

* Determine the maximum tolerated dose (MTD) and clinical response rate for ruxolitinib administered at the higher dose levels.
* Determine safety profile, time to progression
* To test the safety and effectiveness of ruxolitinib for adult T-cell leukemia.

Eligibility:

- Individuals at least 18 years of age who have ATL caused by HTLV-1.

Design:

* Participants will be screened with a physical exam and medical history. Blood and urine samples will be collected. Imaging studies will also be performed.
* Participants will take ruxolitinib twice a day for 28 days. They will have blood tests on days 1, 14, and 28. These tests will look at the levels of HTLV-1 in the blood. Participants will have a final blood test about 2 weeks later. Treatment will also be monitored with imaging studies.
* Participants who have a partial response during treatment may be able to start taking ruxolitinib again after the final blood test. They will continue to take ruxolitinib for as long as it is effective and the side effects are not severe.
* Participants who have a full response during treatment will take ruxolitinib for 56 more days, and then stop treatment. If ATL returns, they may restart treatment and continue it for as long as it is effective.

DETAILED DESCRIPTION:
Background:

* Adult T-cell leukemia is a lymphoproliferative disorder characterized by the presence of cluster of differentiation 4 (CD4)/cluster of differentiation 25 (CD25) expressing T cells (interleukin-2 receptor (IL-2R) alpha expressing) in the peripheral blood, in lymphoid and other tissues.
* In smoldering and chronic adult T-cell leukemia (ATL) the human T-cell leukemia virus 1 (HTLV-1) encoded protein, Tax constitutively activates interleukin-2 (IL-2), IL-9 and IL-15 autocrine/paracrine systems that in turn activate the Janus kinase (JAK)-1/3/signal transducer and activator of transcription 5 (STAT5) pathways.
* Ruxolitinib a therapeutic agent inhibits cytokine mediated Janus kinase (JAK)-1/2 activation and ex vivo proliferation of malignant T cells from subjects with ATL.
* Ruxolitinib is a potent orally bioavailable JAK1/2 inhibitor not licensed for the treatment of ATL.

Primary Objective:

Objective Initial Phase II:

* To determine clinical or objective response rate for ruxolitinib given at 20 mg twice daily
* Primary Objective Dose Escalation Phase I: To determine the maximum tolerated dose and clinical response rate for ruxolitinib given at doses of 30, 40 or 50 mg orally twice daily in subjects with smoldering, chronic and biologically indolent acute or lymphomatous subtype of ATL

Eligibility

* Subjects greater than or equal to 18 years old with pathologically confirmed adult T-cell leukemia: smoldering or chronic or previously treated lymphomatous or acute subtypes with clinically indolent behavior indicated by lack of significant symptoms and treatment free interval of greater than 6 months.
* Subjects must have measurable or evaluable disease. Subjects with > 10% of their PBMCs having the characteristic abnormal (i.e., CD3dim, CD4 plus CD25 plus expressing) fluorescence activated cell sorting (FACS) profile for circulating ATL cells will be considered to have measurable disease.
* Subjects with symptomatic leukemic meningitis, bony or gastrointestinal (GI) tract involvement, serum calcium or Lactate dehydrogenase (LDH) > 1.5 times the upper limit of normal will be excluded. However, subjects that have both ATL and another HTLV-1 associated disease such as tropical spastic paraparesis (human T-cell leukemia virus 1 (HTLV-1) Associated Myelopathy (HAM)/tropical spastic paraparesis (TSP)) will be included.
* No prior treatment with another JAK inhibitor; subjects previously treated in this protocol at the lower dose are eligible to restart treatment at the higher dose levels.

Design

- This is a pilot open-label, trial with off label-use of oral ruxolitinib that will treat 27 to 33 Subjects with smoldering or chronic or clinically indolent ATL. Groups of 3 to 6 newly enrolled or reenrolled Subjects will begin treatment at an elevated dose of 30 mg orally given twice daily. If this dose is tolerated without exceeding the criteria for dose limiting toxicity (DLT) during the first cycle of treatment, the tolerability of treatment at 40 mg and then 50 mg twice daily will be evaluated.

ELIGIBILITY:
* INCLUSION CRITERIA:

NOTE: After approval and activation of Amendment D, subjects who have failed this protocol treatment previously at the initial dose level may be eligible for re-enrollment and retreatment if they otherwise meet eligibility criteria.

* Subjects greater than or equal to 18 years old with pathologically confirmed adult T- cell leukemia: smoldering or chronic, or previously treated lymphomatous or acute subtypes with clinically indolent behavior indicated by lack of significant symptoms and treatment free interval of greater than 6 months are eligible for treatment in the dose escalation and expansion cohorts.
* Subjects must have serum antibodies directed to human T-cell lymphotropic virus type 1 (HTLV-1).
* Subjects must have measurable or evaluable disease. Subjects with > 10% of the peripheral blood mononuclear cells (PBMCs) having the characteristic abnormal (i.e., CD3dim, cluster of differentiation 4 (CD4) plus cluster of differentiation 25 (CD25) plus expressing) fluorescence-activated cell sorting (FACS) profile for circulating adult T-cell leukemia (ATL) cells will be considered to have evaluable disease.
* Subjects must have adequate physiologic parameters:
* Absolute granulocyte count greater than or equal to 500 K/microL, platelet count greater than or equal to 75,000 K/microL and hemoglobin greater than or equal to 10 g/dL.
* Bilirubin and creatinine less than or equal to 1.5 times institutional upper limit of normal (ULN).
* Aspartate aminotransferase (AST), Alanine aminotransferase (ALT) less than or equal to 3.0 times institutional ULN.
* Karnofsky Performance Score greater than or equal to 70% or Eastern Cooperative Oncology Group (ECOG) less than or equal 1.
* Subjects must be able to understand and sign Informed Consent Form.

EXCLUSION CRITERIA:

* Subjects with symptomatic leukemic meningitis, bony or gastrointestinal (GI) tract involvement, serum calcium or lactate dehydrogenase (LDH) > 1.5 times the upper limit of normal will be excluded. However, subjects that have both ATL and another HTLV-1 associated disease such as tropical spastic paraparesis (human T-cell lymphotropic virus type 1 (HTLV-1) Associated Myelopathy (HAM)/tropical spastic paraparesis (TSP) will be included.
* Subjects with symptomatic leukemic meningitis, bony or GI tract involvement, serum calcium or LDH > 1.5 X the upper limit of normal will be excluded. However, subjects that have both ATL and another HTLV-1 associated disease such as tropical spastic paraparesis (HAM/TSP) will be included.
* Subjects who have received high doses of systemic corticosteroids for the treatment of their ATL within 4 weeks prior to the start of therapy.
* Subjects who have received any cytotoxic therapy, immunotherapy, antitumor vaccines or monoclonal antibodies in the 4 weeks prior to the start of the study.
* Life expectancy of less than 3 months.
* Documented active bacterial infections, HTLV-II infection, or hepatitis B or C as follows:

  * A positive hepatitis B serology indicative of previous immunization (i.e., hepatitis B surface antigen (HBsAb) positive and hepatitis B core antibody (HBcAb) negative), or a fully resolved acute hepatitis B infection is not an exclusion criterion.
  * Subjects with an indolent chronic hepatitis B infection (normal ALT, AST, albumin and no radiographic or biopsy evidence of cirrhosis) may be eligible.
  * Subjects with active hepatitis C are excluded. Subjects positive for hepatitis C virus (HCV) antibody are eligible only if polymerase chain reaction (PCR) is negative for HCV ribonucleic acid (RNA).
* Subjects who have untreated human immunodeficiency virus (HIV) are not eligible for this study because by definition they have a defective immune response and are at much higher risk for opportunistic infections due to immune disregulation by both HTLV-1 and HTLVIII (HIV) viruses. Subjects on HIV therapy with undetectable viral loads as measured by HIV RNA quantitative real time PCR may be eligible.
* Inability or refusal to practice effective contraception during therapy. Men and women of childbearing potential must use an effective method of birth control or abstinence during treatment and for 1 week after completion of the treatment.
* Subject has significant and/or uncontrolled cardiac, renal, hepatic or other systemic disorders or significant psychological conditions at baseline visit that in the investigators judgment would jeopardize subject enrollment or compliance with the study procedures.
* Subjects with an absolute requirement for a medication that is a strong inhibitor of Cytochrome P450 3A4 (P450 CYP3A4) are not eligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2012-10-26 (Actual); Primary Completion 2021-11-12 (Actual); Study Completion 2022-01-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin C Conlon, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data (IPD) recorded in the medical record will be shared with intramural investigators upon request.
  All collected IPD will be shared with collaborators under the terms of collaborative agreements.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.
Access Criteria: Clinical data will be made available via subscription to Biomedical Translational Research Information System (BTRIS) and with the permission of the study principal investigator (PI).

REFERENCES:
- [Background] Matsuoka M, Jeang KT. Human T-cell leukemia virus type 1 (HTLV-1) and leukemic transformation: viral infectivity, Tax, HBZ and therapy. Oncogene. 2011 Mar 24;30(12):1379-89. doi: 10.1038/onc.2010.537. Epub 2010 Nov 29. PMID 21119600
- [Background] Tsukasaki K, Hermine O, Bazarbachi A, Ratner L, Ramos JC, Harrington W Jr, O'Mahony D, Janik JE, Bittencourt AL, Taylor GP, Yamaguchi K, Utsunomiya A, Tobinai K, Watanabe T. Definition, prognostic factors, treatment, and response criteria of adult T-cell leukemia-lymphoma: a proposal from an international consensus meeting. J Clin Oncol. 2009 Jan 20;27(3):453-9. doi: 10.1200/JCO.2008.18.2428. Epub 2008 Dec 8. PMID 19064971
- [Background] Yamada Y, Atogami S, Hasegawa H, Kamihira S, Soda M, Satake M, Yamaguchi K. [Nationwide survey of adult T-cell leukemia/lymphoma (ATL) in Japan]. Rinsho Ketsueki. 2011 Nov;52(11):1765-71. Japanese. PMID 22185799
- [Derived] Ohmoto A, Fuji S. Prospects of early therapeutic interventions for indolent adult T-cell leukemia/lymphoma based on the chronic lymphocytic leukemia progression model. Blood Rev. 2023 Jul;60:101057. doi: 10.1016/j.blre.2023.101057. Epub 2023 Feb 20. PMID 36828681
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2013-C-0006.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: No participants were enrolled on dose level 3 or the expansion cohort for the phase I dose escalation version of the protocol because the adult T-cell leukemia (ATL) research program was terminated after the death of the T-cell malignancy group Lead investigator.
Groups:
- Original Phase II Standard Ruxolitinib Dose Cohort - 20 mg Twice Daily: Ruxolitinib 20 mg orally twice daily for 28 days. Subject may continue to receive treatment until progressive disease (PD) or unacceptable toxicity.
- 2- Phase 1 Dose Escalation Cohorts Dose Level 1 - 30 mg Twice Daily: Dose level 1: Ruxolitinib 30 mg orally twice daily for 28 days to determine the maximum tolerated dose (MTD). Subjects may continue to receive treatment until progressive disease (PD) or dose limiting toxicity (DLT) or unacceptable toxicity.
- 2- Phase 1 Dose Escalation Cohorts Dose Level 2 - 40 mg Twice Daily: Dose level 2: Ruxolitinib: Ruxolitinib 40 mg orally twice daily for 28 days to determine the maximum tolerated dose (MTD). Subjects may continue to receive treatment until progressive disease (PD) or dose limiting toxicity (DLT) or unacceptable toxicity.
- 2- Phase 1 Dose Escalation Cohorts Dose Level 3 - 50 mg Twice Daily: Dose level 3: Ruxolitinib: Ruxolitinib 50 mg orally twice daily for 28 days to determine the maximum tolerated dose (MTD). Subjects may continue to receive treatment until progressive disease (PD) or dose limiting toxicity (DLT) or unacceptable toxicity.
Period: Dose Escalation
Arm/Group | Original Phase II Standard Ruxolitinib Dose Cohort - 20 mg Twice Daily | 2- Phase 1 Dose Escalation Cohorts Dose Level 1 - 30 mg Twice Daily | 2- Phase 1 Dose Escalation Cohorts Dose Level 2 - 40 mg Twice Daily | 2- Phase 1 Dose Escalation Cohorts Dose Level 3 - 50 mg Twice Daily | 3- Phase 1 Dose Expansion Cohort
Started | 1 | 5 | 1 | 0 | 0
Completed | 1 | 3 | 1 | 0 | 0
Not Completed | 0 | 2 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 1 | 0 | 0 | 0
Not completed — Unable to take study drug | 0 | 1 | 0 | 0 | 0
Period: Dose Expansion
Arm/Group | Original Phase II Standard Ruxolitinib Dose Cohort - 20 mg Twice Daily | 2- Phase 1 Dose Escalation Cohorts Dose Level 1 - 30 mg Twice Daily | 2- Phase 1 Dose Escalation Cohorts Dose Level 2 - 40 mg Twice Daily | 2- Phase 1 Dose Escalation Cohorts Dose Level 3 - 50 mg Twice Daily | 3- Phase 1 Dose Expansion Cohort
Started | 12 | 0 | 0 | 0 | 0
Completed | 10 | 0 | 0 | 0 | 0
Not Completed | 2 | 0 | 0 | 0 | 0
Not completed — Early disease progression | 1 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 0 | 0
Period: Participants Re-Enrolled and Treated
Arm/Group | Original Phase II Standard Ruxolitinib Dose Cohort - 20 mg Twice Daily | 2- Phase 1 Dose Escalation Cohorts Dose Level 1 - 30 mg Twice Daily | 2- Phase 1 Dose Escalation Cohorts Dose Level 2 - 40 mg Twice Daily | 2- Phase 1 Dose Escalation Cohorts Dose Level 3 - 50 mg Twice Daily | 3- Phase 1 Dose Expansion Cohort
Started | 0 | 1 (Participant treated in the original 20 mg group was re-enrolled and treated at 30 mg twice daily (the protocol allowed this)) | 0 | 0 | 0
Completed | 0 | 1 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Original Phase II Standard Ruxolitinib Dose Cohort - 20 mg Twice Daily | 2- Phase 1 Dose Escalation Cohorts Dose Level 1 - 30 mg Twice Daily | 2- Phase 1 Dose Escalation Cohorts Dose Level 2 - 40 mg Twice Daily | Total
Number analyzed (Participants) | 12 | 6 | 1 | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 10 | 6 | 1 | 17
  >=65 years | 2 | 0 | 0 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.5 (14.5) | 46.3 (10.9) | 65 (0) | 51.93 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 1 | 9
  Male | 7 | 3 | 0 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 12 | 6 | 1 | 19
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 12 | 5 | 1 | 18
  White | 0 | 1 | 0 | 1
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 12 | 6 | 1 | 19
Adult T-Cell Leukemia Lymphoma Diagnosis [Count of Participants; unit: Participants] | 12 | 6 | 1 | 19
Performance Status [Count of Participants; unit: Participants] — Performance status 0 is Normal activity. Fully active, able to carry on all pre-disease performance without restriction. Performance status 1 is symptoms, but ambulatory.
  Restricted in physically strenuous activity, but ambulatory and able to carry out work of a light or sedentary nature (e.g., light housework, office work).
  Participants
    0 | 5 | 4 | 0 | 9
    1 | 7 | 2 | 1 | 10
Prior Therapy [Count of Participants; unit: Participants]
  Surgery | 0 | 0 | 0 | 0
  Chemotherapy | 5 | 3 | 1 | 9
  Radiation Therapy | 5 | 1 | 0 | 6
  Molecular | 0 | 0 | 0 | 0
  Immunotherapy | 5 | 1 | 0 | 6
  Treatment Naive | 4 | 3 | 0 | 7

OUTCOME MEASURES:

1. Primary Outcome: Phase II: Best Response
Description: Best response is complete response (CR) plus partial response (PR). Response was measured by the Revised Response Criteria for Lymphoma by Cheson, et al, and the International Consensus Meeting Criteria for Adult T-Cell Lymphoma (ATL). Complete response is disappearance of all clinical, microscopic, and radiographic evidence of disease. Partial response is a ≥50% reduction in the sum of the products of the greatest diameters of measurable disease without the appearance of new lesion. Stable disease is failure to attain complete response, partial response, or progressive disease. Progressive disease in peripheral blood is defined by a 50% increase from nadir in the count of flower cells and an absolute lymphocyte count, including flower cells, of 4x10^9/L; or the appearance of new lesions excluding skin.
Time Frame: From the time of the start of treatment to approximately 3 years of 5
Measure: Count of Participants; unit: Participants
Arm/Group | Original Phase II Standard Ruxolitinib Dose Cohort - 20 mg Twice Daily | 2- Phase 1 Dose Escalation Cohorts Dose Level 1 - 30 mg Twice Daily | 2- Phase 1 Dose Escalation Cohorts Dose Level 2 - 40 mg Twice Daily
Number analyzed (Participants) | 12 | 6 | 1
Participants
  Complete Response | 0 | 0 | 0
  Partial Response | 1 | 1 | 0
  Stable Disease | 6 | 3 | 0
  Progressive Disease | 5 | 0 | 1
  Not Assessable | 0 | 2 | 0

2. Primary Outcome: Phase I: Maximum Tolerated Dose (MTD)
Description: MTD is defined as the dose level at which no more than 1 of up to 6 participants experience dose-limiting toxicity (DLT) during the first cycle (28 days) treatment, and the dose below that at which at least 2 (of ≤6) participants have DLT as a result of the drug. A DLT is any grade 3 or 4 toxicity, if deemed possibly, probably, or definitely related to the study drug by the principal investigator during the first cycle of treatment with some exceptions such as Grade 3 anemia without hemolysis. Grade 3 or 4 granulocytopenia or leukopenia without infection, Grade 3 thrombocytopenia without bleeding, and Grade 3 or 4 lymphopenia. Grade 3 is severe or medically significant. Grade 4 is life-threatening, urgent intervention indicated.
Time Frame: From the time of the start of treatment to approximately 1 year
Population: No participants were treated in an expansion cohort (50mg) before the protocol was closed.
Measure: Number; unit: mg
Arm/Group | 2- Phase 1 Dose Escalation Cohorts Dose Level 1 - 30 mg Twice Daily | 2- Phase 1 Dose Escalation Cohorts Dose Level 2 - 40 mg Twice Daily | 2- Phase 1 Dose Escalation Cohorts Dose Level 3 - 50 mg Twice Daily
Number analyzed (Participants) | 6 | 1 | 0
mg | NA — MTD was not defined because the Adult T-Cell Leukemia (ATL) project was terminated. | NA — MTD was not defined because the Adult T-Cell Leukemia (ATL) project was terminated. |

3. Secondary Outcome: Phase II: Time to Progression (TTP)
Description: TTP is defined as the date of protocol consent until date of progressive disease is documented. Progressive disease was assessed by the Revised Response Criteria for Lymphoma by Cheson, et al, and the International Consensus Meeting Criteria for Adult T-Cell Lymphoma (guideline (version 1.1). Progressive disease (PD) is at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study, and the appearance of one or more new lesions.
Time Frame: From the time of the start of treatment to approximately 3 years
Measure: Mean (Standard Deviation); unit: Months
Arm/Group | Original Phase II Standard Ruxolitinib Dose Cohort - 20 mg Twice Daily | 2- Phase 1 Dose Escalation Cohorts Dose Level 1 - 30 mg Twice Daily | 2- Phase 1 Dose Escalation Cohorts Dose Level 2 - 40 mg Twice Daily
Number analyzed (Participants) | 12 | 5 | 1
Months | 5.25 (7.62) | 3.36 (3.34) | 1 (NA) — Standard deviation is NA because it is only one participant.

4. Secondary Outcome: Phase II: Survival Time
Description: Survival time is defined as the date of protocol consent until the date of the subject's death for any cause.
Time Frame: From the time of the start of treatment to approximately 3 years
Measure: Mean (95% Confidence Interval); unit: Months
Arm/Group | Original Phase II Standard Ruxolitinib Dose Cohort - 20 mg Twice Daily | 2- Phase 1 Dose Escalation Cohorts Dose Level 1 - 30 mg Twice Daily | 2- Phase 1 Dose Escalation Cohorts Dose Level 2 - 40 mg Twice Daily
Number analyzed (Participants) | 12 | 6 | 1
Months | 29.3 [15.7 to 42.9] | 20.1 [3.9 to 36.3] | 14.1 [NA to NA] — 95% confidence interval cannot be calculated for one participant.

5. Secondary Outcome: Phase I: Grade of Serious and/or Non-serious Adverse Events (SAEs) Related to the Experimental Treatment by Grade
Description: Grade of serious adverse events (SAEs) related to the experimental treatment. Adverse events were assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0). Grade 1 is mild, Grade 2 is moderate, Grade 3 is severe, and Grade 4 is life-threatening.
Time Frame: From the time of the start of treatment to approximately 1 year
Measure: Number; unit: Adverse Events
Groups:
- Grade 1 - Original Phase II Standard Ruxolitinib Dose Cohort - 20 mg Twice Daily; Grade 2 - Original Phase II Standard Ruxolitinib Dose Cohort - 20 mg Twice Daily; Grade 3 - Original Phase II Standard Ruxolitinib Dose Cohort - 20 mg Twice Daily; Grade 4 - Original Phase II Standard Ruxolitinib Dose Cohort - 20 mg Twice Daily: Ruxolitinib 20 mg orally twice daily for 28 days. Subject may continue to receive treatment until progressive disease (PD) or unacceptable toxicity.
- Grade 1 - 2- Phase 1 Dose Escalation Cohorts Dose Level 1 - 30 mg Twice Daily; Grade 2 - Phase 1 Dose Escalation Cohorts Dose Level 1 - 30 mg Twice Daily; Grade 3 - Phase 1 Dose Escalation Cohorts Dose Level 1 - 30 mg Twice Daily; Grade 4 - Phase 1 Dose Escalation Cohorts Dose Level 1 - 30 mg Twice Daily: Dose level 1: Ruxolitinib 30 mg orally twice daily for 28 days to determine the maximum tolerated dose (MTD). Subjects may continue to receive treatment until progressive disease (PD) or dose limiting toxicity (DLT) or unacceptable toxicity.
- Grade 1 - 2- Phase 1 Dose Escalation Cohorts Dose Level 2 - 40 mg Twice Daily; Grade 2 - 2- Phase 1 Dose Escalation Cohorts Dose Level 2 - 40 mg Twice Daily; Grade 3 - 2- Phase 1 Dose Escalation Cohorts Dose Level 2 - 40 mg Twice Daily; Grade 4 - 2- Phase 1 Dose Escalation Cohorts Dose Level 2 - 40 mg Twice Daily: Dose level 2: Ruxolitinib: Ruxolitinib 40 mg orally twice daily for 28 days to determine the maximum tolerated dose (MTD). Subjects may continue to receive treatment until progressive disease (PD) or dose limiting toxicity (DLT) or unacceptable toxicity.
Arm/Group | Grade 1 - Original Phase II Standard Ruxolitinib Dose Cohort - 20 mg Twice Daily | Grade 2 - Original Phase II Standard Ruxolitinib Dose Cohort - 20 mg Twice Daily | Grade 3 - Original Phase II Standard Ruxolitinib Dose Cohort - 20 mg Twice Daily | Grade 4 - Original Phase II Standard Ruxolitinib Dose Cohort - 20 mg Twice Daily | Grade 1 - 2- Phase 1 Dose Escalation Cohorts Dose Level 1 - 30 mg Twice Daily | Grade 2 - Phase 1 Dose Escalation Cohorts Dose Level 1 - 30 mg Twice Daily | Grade 3 - Phase 1 Dose Escalation Cohorts Dose Level 1 - 30 mg Twice Daily | Grade 4 - Phase 1 Dose Escalation Cohorts Dose Level 1 - 30 mg Twice Daily | Grade 1 - 2- Phase 1 Dose Escalation Cohorts Dose Level 2 - 40 mg Twice Daily | Grade 2 - 2- Phase 1 Dose Escalation Cohorts Dose Level 2 - 40 mg Twice Daily | Grade 3 - 2- Phase 1 Dose Escalation Cohorts Dose Level 2 - 40 mg Twice Daily | Grade 4 - 2- Phase 1 Dose Escalation Cohorts Dose Level 2 - 40 mg Twice Daily
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 6 | 6 | 6 | 6 | 1 | 1 | 1 | 1
Adverse Events
  Fatigue | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Nausea | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Anemia | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Alanine aminotransferase increased | 3 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Aspartate aminotransferase increased | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocyte count decreased | 3 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Bilirubin increased | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White blood cells decreased | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Platelet count decreased | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Creatinine increased | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypernatremia | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Alkaline phosphatase increased | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophil count decreased | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0

6. Secondary Outcome: Phase I: Time to Progression When Ruxolitinib is Administered at Doses of 30, 40 or 50 mg Orally Twice Daily
Description: TTP is defined as the date of protocol consent until date of progressive disease is documented. Progressive disease was assessed by the Revised Response Criteria for Lymphoma by Cheson, et al, and the International Consensus Meeting Criteria for Adult T-Cell Lymphoma guidelines (version 1.1). Progressive disease (PD) is at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study, and the appearance of one or more new lesions.
Time Frame: From the time of the start of treatment to approximately 1 year
Population: No participants were enrolled on the expansion cohort for the phase I dose escalation (50mg) version of the protocol.
Measure: Mean (95% Confidence Interval); unit: Months
Arm/Group | Original Phase II Standard Ruxolitinib Dose Cohort - 20 mg Twice Daily | 2- Phase 1 Dose Escalation Cohorts Dose Level 1 - 30 mg Twice Daily | 2- Phase 1 Dose Escalation Cohorts Dose Level 2 - 40 mg Twice Daily | 2- Phase 1 Dose Escalation Cohorts Dose Level 3 - 50 mg Twice Daily
Number analyzed (Participants) | 12 | 6 | 1 | 0
Months | 5.2 [0.89 to 9.51] | 4.1 [0.77 to 7.43] | 1 [NA to NA] — 95% confidence interval cannot be calculated for one participant. |

7. Other Pre Specified Outcome: Number of Participants With a Dose Limiting Toxicity (DLT)
Description: A DLT is any grade 3 or 4 toxicity, if deemed possibly, probably or definitely related to the study drug by the principal investigator during the first cycle of treatment with some exceptions such as Grade 3 anemia without hemolysis. Grade 3 or 4 granulocytopenia or leukopenia without infection, Grade 3 thrombocytopenia without bleeding, and Grade 3 or 4 lymphopenia. Grade 3 is severe or medically significant. Grade 4 is life-threatening, urgent intervention indicated.
Time Frame: During the first cycle of treatment (28 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Original Phase II Standard Ruxolitinib Dose Cohort - 20 mg Twice Daily | 2- Phase 1 Dose Escalation Cohorts Dose Level 1 - 30 mg Twice Daily | 2- Phase 1 Dose Escalation Cohorts Dose Level 2 - 40 mg Twice Daily
Number analyzed (Participants) | 12 | 6 | 1
Participants | 0 | 0 | 0

8. Other Pre Specified Outcome: Number of Participants With Non-Serious Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0).
Description: Here is the number of participants with non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0). A non-serious adverse event is any untoward medical occurrence.
Time Frame: Date treatment consent signed to date off study, approximately 110 months and 27 days.
Measure: Count of Participants; unit: Participants
Arm/Group | Original Phase II Standard Ruxolitinib Dose Cohort - 20 mg Twice Daily | 2- Phase 1 Dose Escalation Cohorts Dose Level 1 - 30 mg Twice Daily | 2- Phase 1 Dose Escalation Cohorts Dose Level 2 - 40 mg Twice Daily
Number analyzed (Participants) | 12 | 6 | 1
Participants | 12 | 6 | 1

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 110 months and 27 days.
Arm/Group | Original Phase II Standard Ruxolitinib Dose Cohort - 20 mg Twice Daily | 2- Phase 1 Dose Escalation Cohorts Dose Level 1 - 30 mg Twice Daily | 2- Phase 1 Dose Escalation Cohorts Dose Level 2 - 40 mg Twice Daily
All-Cause Mortality (participants affected / at risk) | 11/12 | 3/6 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/6 | 0/1
Other Adverse Events (participants affected / at risk) | 12/12 | 6/6 | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Original Phase II Standard Ruxolitinib Dose Cohort - 20 mg Twice Daily (N=12) | 2- Phase 1 Dose Escalation Cohorts Dose Level 1 - 30 mg Twice Daily (N=6) | 2- Phase 1 Dose Escalation Cohorts Dose Level 2 - 40 mg Twice Daily (N=1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 3 (5) | 2 (2) | 0 (0)
Alkaline phosphatase increased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 3 (7) | 1 (1) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 3 (5) | 1 (1) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Creatinine increased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Edema limbs (General disorders) | 2 (2) | 0 (0) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0)
Fever (General disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (4) | 0 (0) | 0 (0)
Infections and infestations - Other, Chikungunya virus (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infections and infestations - Other, Haemophilus influenzae bacteremia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infections and infestations - Other, Shingles (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Infusion site extravasation (General disorders) | 1 (1) | 0 (0) | 0 (0)
Investigations - Other, Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 7 (10) | 2 (3) | 0 (0)
Lymphocyte count increased (Investigations) | 1 (1) | 1 (2) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 6 (9) | 3 (3) | 1 (6)
Pain (General disorders) | 4 (4) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Paresthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 2 (2) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Serum amylase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - Other, callous buildup on toes (unsure if related to ATL) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
White blood cell decreased (Investigations) | 7 (7) | 0 (0) | 1 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-02-10): https://cdn.clinicaltrials.gov/large-docs/59/NCT01712659/Prot_SAP_000.pdf
  • Informed Consent Form (2021-01-11): https://cdn.clinicaltrials.gov/large-docs/59/NCT01712659/ICF_001.pdf